CLINICAL TRIAL: NCT04456842
Title: Cardiovascular Registry of Atrial Fibrillation in Latin America: The LACROSS Study
Brief Title: Cardiovascular Registry of Atrial Fibrillation
Acronym: LACROSS
Status: Completed | Type: Observational
Sponsor: Brazilian Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 001/2018
Record Dates: First submitted 2020-06-23; First posted 2020-07-07 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrilation; Antithrombotic therapy; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient Registry Data — To set data on demographic characteristics,documenting antithrombotic therapy, describe the INR control level of VKA users, discontinuation rates and clinical outcomes, such as stroke, hemorrhage and death.

SUMMARY:
Follow a representative sample of Latin American patients diagnosed with atrial fibrillation to set data on demographic characteristics, documenting antithrombotic therapy, describe the INR control level of VKA users, discontinuation rates and clinical outcomes, such as stroke, hemorrhage and death

DETAILED DESCRIPTION:
Patients will be followed 6 months and 1 year after the baseline visit and will be collected data of antithrombotic therapy, laboratory data, discontinuation rates of antithrombotic therapy and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years-old that signed informed consent;
* Atrial Fibrillation or Atrial Flutter at the time of inclusion documented in source document;
* If the patient is not in atrial fibrillation or Atrial Flutter rhythm, s/he should have 2 electrographic records, at least 15 days apart between them, with one of them being performed within the last 6 months before enrollment (AF may be documented by 12-lead ECG, Holter monitor-24h);

Exclusion Criteria:

* Patients who did not agree to participate.
* Patients without possibility of monitoring for one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Atrial Fibrilation or Atrial Flutter
Sampling Method: Probability Sample
Enrollment: 2016 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
INR control rate | 12 months
Oral anticoagulation discontinuation rate | 12 months
Percentage of death | 12 months
Percentage of stroke | 12 months
Percentage of systemic embolism | 12 months
Percentage of myocardial infarction | 12 months
Percentage of major bleeding | 12 months
Percentage of electrical cardioversion | 12 months
Percentage of percutaneous ablation of AF | 12 months
Percentage of atrioventricular junction ablation | 12 months
Percentage of patients that need of pacemaker implantation | 12 monts
Percentage of other cardiovascular hospitalization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renato D. Lopes, MD, PhD, Study Chair — Instituto Brasileiro de Pesquisa Thomaz de Carvalho - BCRI
Locations (17):
- Argentina (11):
  - Hospital Interzonal General de Agudos "Dr. José Penna", Bahía Blanca, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Centro de Investigaciones Medicas Temperley (CIMeT), Temperley, Buenos Aires
  - Hospital Italiano de La Plata, Buenos Aires, La Plata
  - Centro Modelo de Cardiologia, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Luquez, Córdoba
  - Prevención Cardiovascular Salta, Salta
  - Servicios Médicos El Castaño, San Juan
  - Instituto Cardiovascular San Luis, San Luis
  - Centro de Investigaciones Clinicas del Litoral SRL, Santa Fe
  - Hospital Provincial Dr. José Maria Cullen, Santa Fe
- Hospital Alvorada Taguatinga Ltda, São Paulo, Brazil
- Colombia (2):
  - Sociedad de Cirugia de Bogota - Hospital de San Jose, Bogotá, Cundinamarca
  - Fundacion Valle del Lili, Cali, Valle del Cauca Department
- Mexico (3):
  - Francisco Gerardo Padilla Padilla, Guadalajara, Jalisco
  - Centro de Estudios Clínicos de Queretaro S.C. (CECLIQ), Querétaro City, Querétaro
  - Centro para el Desarrollo de la Medicina y de Asistecia Medica Especializada S.C., Culiacán, Sinaloa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR